CLINICAL TRIAL: NCT05861869
Title: Clinical Trial of PLA2R-IgG4 Detection Kit (Time-resolved Fluorescence Immunoassay)
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Zhejiang Biostar Biotechnology Co. (Industry)
Collaborators: First Affiliated Hospital of Zhejiang University (Other); Wuxi People's Hospital (Other); Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZJBS-PLA2R IgG4-2201
Record Dates: First submitted 2023-04-10; First posted 2023-05-17 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2023-05

CONDITIONS: Membranous Nephropathy - PLA2R Induced; Kidney Diseases-except Membranous Nephropathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PLA2R-induced membranous nephropathy group: 1. Pathological examination showed that patients with membranous nephropathy were positive for PLA2R by immunohistochemistry, and the symptoms were not completely relieved; (24 h urine protein quantification<0.3g or urine protein /creatinine (uPCR)<300mg /g is regarded as complete remission)
  2. In patients with nephrotic syndrome (serum albumin ≤ 30.0g /L, clinical manifestations show moderate to large amount of proteinuria (urine protein>3.5g /L or urine protein /creatinine ratio ≥ 3500mg /g), and their serum anti PLA2R antibody detection shows positive.
- Secondary membranous nephropathy group: 1. Patients in nephrology department who have ruled out primary membranous nephropathy.
  2. the patient has the remaining serum samples of normal test, and the serum volume of the sample is not less than 1ml.

SUMMARY:
The goal of this observational clinical trial is to compare assessment reagents with clinical diagnostic criteria in patients with membranous nephropathy. The main questions it aims to answer are:

* Evaluating the sensitivity and specificity of the test reagent in the diagnosis of membranous nephropathy.
* Evaluating whether the clinical diagnostic performance of the test reagent meets the requirements for auxiliary diagnosis of membranous nephropathy.

Participants will provide approximately 4ml of blood. Researchers will compare the levels of anti-PLA2RIgG4 in patients with membranous nephropathy and patients with other renal diseases,to see if there is a significant difference.

ELIGIBILITY:
Inclusion Criteria:

* PLA2R-induced membranous nephropathy group

  1. Pathological examination showed that patients with membranous nephropathy were positive for PLA2R by immunohistochemistry, and the symptoms were not completely relieved; (24 h urine protein quantification<0.3g or urine protein /creatinine (uPCR)<300mg /g is regarded as complete remission)
  2. In patients with nephrotic syndrome (serum albumin ≤ 30.0g /L, clinical manifestations show moderate to large amount of proteinuria (urine protein>3.5g /L or urine protein /creatinine ratio ≥ 3500mg /g), and their serum anti PLA2R antibody detection shows positive.
* Secondary membranous nephropathy group Patients in nephrology department who have ruled out primary membranous nephropathy.

the patient has the remaining serum samples of normal test, and the serum volume of the sample is not less than 1ml.

Exclusion Criteria:

1. The amount of centrifuged serum sample after blood collection is less than 1ml or the amount of residual serum in normal test is less than 1ml;
2. Non-serum samples, plasma samples;
3. Patients with mental or cognitive disorders;
4. No samples with definite clinical diagnosis;
5. Samples with incomplete information.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Nephrology department visit /inpatient case
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Content of anti-PLA2r IgG4 | through study completion, an average of 1 year
  Evaluating the sensitivity and specificity of the test reagent in the diagnosis of membranous nephropathy

CONTACTS AND LOCATIONS:
Locations (1):
- ZhejiangBiostar, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No